CLINICAL TRIAL: NCT00844519
Title: Effect of Maraviroc on Endothelial Function in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIVCADRFA
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infection; Cardiovascular Disease; Inflammation; HIV Infections
Keywords: Treatment Experienced; CCR5 receptor; maraviroc
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases; Inflammation; Diabetes Mellitus, Insulin-Dependent, 22 | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Active Comparator): For subjects assigned to the maraviroc group, subjects will receive maraviroc at 300mg by mouth twice daily for 24 weeks in addition to taking their current anti-HIV medication. For subjects on ritonavir, the dose of maraviroc will be 150mg by mouth twice daily.
  Interventions: Drug: Maraviroc
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Maraviroc — For subjects assigned to the maraviroc group, they will receive maraviroc at 300mg by mouth twice daily for 24 weeks in addition to taking their current anti-HIV medications. For subjects on ritonavir, the dose will be reduced to 150mg by mouth twice daily for 24 weeks.
  Arms: Maraviroc
Drug: placebo — For subjects assigned to the placebo group, they will receive a matching placebo pill 300mg to be taken by mouth twice daily for 24 weeks in addition to taking their current anti-HIV medications.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the potentially beneficial aspects of CCR5 inhibition on inflammation and endothelial function as measured by brachial artery reactivity in antiretroviral treated HIV patients with an undetectable viral load.

ELIGIBILITY:
Inclusion Criteria:

1. Stable antiretroviral therapy for at least 12 months
2. All plasma HIV RNA levels within the past year must be below level of detection (< 50 copies RNA/mL), although isolated single values > 50 but < 200 copies will be allowed.
3. Screening plasma HIV RNA levels < 50 copies RNA/mL
4. >90% adherence to therapy within the preceding 30 days, as determined by self-report
5. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.

Exclusion Criteria:

1. Ongoing or prior use of any integrase inhibitor or R5 inhibitor.
2. Patients who plan to modify existing antiretroviral therapy in the next 24 weeks for any reason
3. Serious illness requiring hospitalization or parental antibiotics within preceding 3 months
4. Concurrent or recent exposure to any immunomodulatory drugs
5. Advanced liver disease or active hepatitis B or C
6. Patients with systolic blood pressure <100/70
7. Starting or stopping statin therapy during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc: maraviroc at 300mg by mouth twice daily for 24 weeks in addition to current anti-HIV medication regimen. For subjects on ritonavir, the dose of maraviroc will be 150mg by mouth twice daily.
- Placebo: matching placebo pill 300mg by mouth twice daily for 24 weeks in addition to current anti-HIV medication regimen.
Period: Overall Study
Arm/Group | Maraviroc | Placebo
Started | 26 | 26
Completed | 24 | 25
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: per protocol
Groups:
- Maraviroc: maraviroc at 300mg by mouth twice daily for 24 weeks in addition to current anti-HIV medication regimen. For subjects on ritonavir, the dose of maraviroc was 150mg by mouth twice daily.
- Total: Total of all reporting groups
Arm/Group | Maraviroc | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [45 to 60] | 52 [47 to 57] | 52 [45 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 25 | 26 | 51
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in FMD
Description: endothelial function as assessed by measured flow-mediated vasodilation (FMD) of the brachial artery
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: percent change in FMD
Groups:
- Maraviroc: maraviroc 300mg by mouth twice daily for 24 weeks in addition to current anti-HIV medication regimen. For subjects on ritonavir, the dose of maraviroc was 150mg by mouth twice daily.
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 26 | 26
percent change in FMD | 0.57 (2.1) | -0.05 (2.1)
Statistical Analysis 1: Comparison: Maraviroc; within-arm, pre-post change in FMD; Test type: Superiority or Other; p = 0.17, t-test, 2 sided — significant at p<0.05
Statistical Analysis 2: Comparison: Placebo; within-arm, pre-post change in FMD; Test type: Superiority or Other; p = 0.90, t-test, 2 sided — significant at p<0.05

ADVERSE EVENTS:
Arm/Group | Maraviroc | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=26) | Placebo (N=26)
hepatocellular carcinoma (Surgical and medical procedures) | 1 (1) | 0 (0) — Small mass found at ultrasound, later determined to be hepatocellular carcinoma. It is unlikely that this mass is a result of the study medication, as the patient had only been on the medication for 14 days when mass was found at ultrasound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No